CLINICAL TRIAL: NCT04334954
Title: SARS-COV2 Pandemic Serosurvey and Blood Sampling
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200083; 20-I-0083
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: SARS-COV2 Virus
Keywords: COVID-19; Immunity; Antibodies; Respiratory Virus; Virus; Natural History
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers

SUMMARY:
Background:

Respiratory virus outbreaks and pandemics, such as SARS, MERS, and the new SARS-COV2 virus, have major impacts worldwide. Researchers must act quickly to learn about the exposures and immunity in the general population. This can be done by studying people s blood serum to find those with antibodies to the virus. This knowledge can help in current and future pandemics. In this study, researchers want to find people who have anti-SARS-COV2 antibodies but no known exposure or illness.

Objective:

To find the number of people with detectable antibodies to SARS-COV2 from a sampling of adults who have no known exposure or clinical illness.

Eligibility:

Adults ages 18 and older without a confirmed COVID19 infection or current symptoms consistent with COVID19

Design:

Participants will enroll and give consent over the phone. They will be screened over the phone with a health assessment questionnaire. They will be screened for COVID19 using the NIH COVID19 screening questionnaire.

Participants will give a blood sample. They can go to the NIH Clinical Center or do home blood sampling. In-person collection at NIH is preferred.

If participants go to NIH, 2 tubes of blood will be taken.

If participants do home sampling, they will be sent a home sampling kit. The kit contains gauze, an alcohol pad, a lancet, collection devices, and shipping materials. It also contains detailed instructions. They will collect 80ul of blood and mail it to the NIH lab.

Participants may enroll in the study up to 4 times. They cannot enroll within 30 days of previous enrollment.

DETAILED DESCRIPTION:
It has been demonstrated that respiratory virus outbreaks and pandemics, such as influenza, SARS, MERS, and now the newly emerged SARS-COV2 virus, have a major impact on morbidity and mortality worldwide, as well as having devastating global economic and societal impact. During these outbreaks it is critical to gain a rapid understanding of the exposures and immunity in the general population. Identifying exposures can be accomplished through analysis of serum during an outbreak to identify those with specific antibodies to the pathogen. The knowledge of the level of exposures could greatly impact the response to current and future pandemics. In this natural history study, we will collect blood from individuals to identify those who have anti-SARS-COV2 antibodies present despite no confirmed disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. >= 18 years of age.
  2. Willing and able to complete a verbal telephone consent.
  3. Willing to undergo one blood draw or home blood sampling.
  4. Willing to have blood samples stored for future research.
  5. Have previously participated in Phase 1 of this study (inclusion for Phase II only)

Co-enrollment Guidelines

Participants may be co-enrolled in other research studies.

EXCLUSION CRITERIA:

1. Confirmed history of COVID19 infection or exposure (exclusion for Phase I only)
2. Current symptoms consistent with COVID19 infection
3. Any condition or event that, in the PI s opinion, may substantially increase the risk associated with study participation or compromise the study's scientific objectives. Conditions that exclude a subject are considered to be unlikely, but an example would include having a blood clotting disorder that would make it unsafe to obtain blood samples.
4. Not willing to have blood samples stored for future research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 11363 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Number of people with detectable antibodies to SARS-COV2 and follow them over one year to evaluate change over a 12 month period | 2 years
  Anti-SARS-COV2 IgG and IgM ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
.Data will be shared per existing DUA with RDCRN and study sites. @@@@@@Unidentifiable IPD will also be made public through NCI seronet.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be shared starting a maximum of 1 year after publication.
Access Criteria: The IPD will be available publicly.

REFERENCES:
- [Derived] Kalish H, Klumpp-Thomas C, Hunsberger S, Baus HA, Fay MP, Siripong N, Wang J, Hicks J, Mehalko J, Travers J, Drew M, Pauly K, Spathies J, Ngo T, Adusei KM, Karkanitsa M, Croker JA, Li Y, Graubard BI, Czajkowski L, Belliveau O, Chairez C, Snead K, Frank P, Shunmugavel A, Han A, Giurgea LT, Rosas LA, Bean R, Athota R, Cervantes-Medina A, Gouzoulis M, Heffelfinger B, Valenti S, Caldararo R, Kolberg MM, Kelly A, Simon R, Shafiq S, Wall V, Reed S, Ford EW, Lokwani R, Denson JP, Messing S, Michael SG, Gillette W, Kimberly RP, Reis SE, Hall MD, Esposito D, Memoli MJ, Sadtler K. Mapping a Pandemic: SARS-CoV-2 Seropositivity in the United States. medRxiv [Preprint]. 2021 Jan 31:2021.01.27.21250570. doi: 10.1101/2021.01.27.21250570. PMID 33532807
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0083.html